CLINICAL TRIAL: NCT01591941
Title: The Effectiveness of a Novel Warm-up in Decreasing Risk Factors for Anterior Cruciate Ligament Injury in Female Youth Soccer Players
Brief Title: Effectiveness of a Novel Warm-up in Decreasing Risk Factors for ACL Injury in Female Youth Soccer Players
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BCM06-0007
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: ACL Injury
Keywords: ACL, Knee , Injury,
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CON group (Active Comparator): Control Group underwent a standard soccer warm-up
  Interventions: Other: Core-PAC
- Core-PAC (Experimental): Experimental took part in the Core position and control movement strategy (Core-PAC) warm-up
  Interventions: Other: Core-PAC

INTERVENTIONS:
Other: Core-PAC — Core position and control movement strategy (Core-PAC):
  Do warm-up prior to 6 weeks of regular soccer training for peak flexion angles and peak abduction moments at the knee during a side-cut (SC) and an unanticipated side-cut (USC) prior to kicking a soccer ball and a side-hop (SH) task.

SUMMARY:
There is a large number of young women who sustain serious knee injuries from playing soccer. Female athletes are at high risk of knee injuries from soccer than males. We will conduct a research project to assess the effect of a warm-up on changing some of the movement patterns thought to contribute to these serious knee injuries.

It is hypothesized that a core position and control movement strategy (Core-PAC) group reduce biomechanical risk factors at the knee compared to a control after the training program.

DETAILED DESCRIPTION:
There is a large number of young women who sustain serious knee injuries from playing soccer. Female athletes are at high risk of knee injuries from soccer than males. We will conduct a research project to assess the effect of a warm-up on changing some of the movement patterns thought to contribute to these serious knee injuries.

A core position and control movement strategy (Core-PAC) may be one method of modifying high-risk movements such as side-cutting. The Core-PAC is a simple method of getting the centre of mass (COM) closer to the plant foot or base of support (BOS). Moving the COM closer to the BOS may bias joint loading to the sagittal rather than the frontal and transverse planes, which often occurs in female athletes and poses a risk for ACL injury.

In this study, we will conduct a randomized controlled trial to compare a Core-PAC trained group to a control group for peak flexion angles and peak abduction moments at the knee during a side-cut and an unanticipated side-cut prior to kicking a soccer ball and a side-hop task after a six-week training program.

It is hypothesized that a Core-PAC group would have greater peak flexion angles and lower peak abduction moments at the knee compared to a control after the training program.

ELIGIBILITY:
Inclusion Criteria:

* 14-17 years of age;
* have no injuries for six weeks prior to testing;
* have no medical problems preventing them from participating in the study.

Exclusion Criteria:

* have a previous ACL injury or repair;
* have a back or lower limb injury that kept them from playing or training for greater than 30 days in the past year;
* presently using a supplemental exercise based program;
* have any medical or neurologic condition that would impair their ability to perform the tasks.

Ages: 14 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Peak knee flexion angle and peak abduction moment | 6 weeks
  Intervention group will be instructed to move from the trunk first during a series of athletic tasks. The Control group will be instructed to move with their usual athletic movements during the same tasks.
  After 6 weeks of this training, subjects will be asked to return to the GF Strong Rehabilitation Center for biomechanical testing.

CONTACTS AND LOCATIONS:
Overall Officials: Suan R Harris, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Rehab Research Lab, GF Strong Rehab Centre, Vancovuer, British Columbia, Canada